CLINICAL TRIAL: NCT03079531
Title: An Open Label Phase 1b Study of Secukinumab in Patients With Moderate to Severe Papulopustular Rosacea
Brief Title: Open Label Study to Assess the Effect of Secukinumab in Moderate to Severe Papulopustular Rosacea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Anne Chang (Other)
Responsible Party: Sponsor-Investigator, Anne Chang, Associate Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-protocol 38599
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Papulopustular Rosacea
MeSH Terms: conditions — Rosacea | interventions — secukinumab; guselkumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Secukinumab arm (Experimental): Participants receive secukinumab (7 doses over a 16-week study period).
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab 300 mg administered subcutaneously.
  Other Names: Tremfya

SUMMARY:
This is a study to determine whether secukinumab is a potential therapy for those with papulopustular rosacea. We will observe whether this drug decreases the size and/or amount and severity of the pustules of those who suffer from rosacea.

DETAILED DESCRIPTION:
Rosacea is a common inflammatory skin disease affecting up to 10% of adults. Despite this, the etiology of rosacea is unclear, although there may be a genetic predisposition (Chang et al., 2015). Currently, there is no cure. Rosacea can lead to scarring, itching, burning, and is associated with anxiety and depression (Moustafa et al., 2015), significantly affecting quality of life.

Secukinumab is an antibody that binds to a protein (interleukin (IL)-17A) that is involved in inflammation. When IL-17A is bound to secukinumab, it cannot bind to its receptor, thereby inhibiting its ability to feed the inflammatory response. In clinical trials, secukinumab has been effective for moderate to severe psoriasis (Blauvelt et al., 2015). Recently, human data from all types of rosacea have shown Th1/Th17 polarization profile of the T-cell response, suggesting that anti-IL-17 therapy may be beneficial for rosacea (Buhl et al., 2015). Hence, secukinumab could be effective against rosacea. This proposal is a proof-of-concept study to use secukinumab in open label design for moderate to severe papulopustular rosacea.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe papulopustular rosacea defined clinically using the grading system of Wilkin et al. (2004) as having at least ten lesions (either papules or pustules) on face at time of enrollment
* age 18 years or greater willing and able to understand and sign informed consent form

Exclusion Criteria:

* known hypersensitivity to secukinumab
* topical or oral anti-rosacea medication usage for 28 days prior to enrollment
* active Crohn's disease, as secukinumab may exacerbate this disease
* active infection including tuberculosis, hepatitis B or C, human immunodeficiency virus
* participants with latent tuberculosis will need to have treatment initiated prior to starting study drug
* pregnant or lactating
* active and/or uncontrolled medical conditions that may interfere with study procedures or obscure rosacea assessment such as cutaneous lupus
* use of retinoids within past 3 months of enrollment
* use of antibiotics within 4 weeks of enrollment
* use of light based or laser treatment to face within 8 weeks of enrollment
* use of topical or systemic steroids within 4 weeks of enrollment
* acne conglobate, acne fulminans, chloracne, severe acne requiring systemic treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Chang, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Dermatology, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang ALS, Raber I, Xu J, Li R, Spitale R, Chen J, Kiefer AK, Tian C, Eriksson NK, Hinds DA, Tung JY. Assessment of the genetic basis of rosacea by genome-wide association study. J Invest Dermatol. 2015 Jun;135(6):1548-1555. doi: 10.1038/jid.2015.53. Epub 2015 Feb 19. PMID 25695682
- [Background] Moustafa F, Hopkinson D, Huang KE, Feldman S. Prevalence of rosacea in community settings. J Cutan Med Surg. 2015 Mar-Apr;19(2):149-52. doi: 10.2310/7750.2014.14087. Epub 2015 Mar 11. PMID 25775639
- [Background] Blauvelt A, Prinz JC, Gottlieb AB, Kingo K, Sofen H, Ruer-Mulard M, Singh V, Pathan R, Papavassilis C, Cooper S; FEATURE Study Group. Secukinumab administration by pre-filled syringe: efficacy, safety and usability results from a randomized controlled trial in psoriasis (FEATURE). Br J Dermatol. 2015 Feb;172(2):484-93. doi: 10.1111/bjd.13348. Epub 2014 Dec 11. PMID 25132411
- [Background] Buhl T, Sulk M, Nowak P, Buddenkotte J, McDonald I, Aubert J, Carlavan I, Deret S, Reiniche P, Rivier M, Voegel JJ, Steinhoff M. Molecular and Morphological Characterization of Inflammatory Infiltrate in Rosacea Reveals Activation of Th1/Th17 Pathways. J Invest Dermatol. 2015 Sep;135(9):2198-2208. doi: 10.1038/jid.2015.141. Epub 2015 Apr 7. PMID 25848978

RESULTS

PARTICIPANT FLOW:
Groups:
- Secukinumab Arm: Secukinumab 300 mg administered subcutaneously (7 doses over a 16-week study period).
Period: Overall Study
Arm/Group | Secukinumab Arm
Started | 24
Attended ≥1 Post-baseline Visit | 23
Completed | 17
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: Participants with at least one post-baseline visit were considered evaluable in this trial, and are included in the analysis for Baseline Characteristics.
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 23
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56 [50 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 18
  Black | 1
  Hispanic/Latino | 2
  Asian | 1
  Two or More Races | 1
Region of Enrollment [Number; unit: participants]
  United States | 23
Papule/pustule count [Median (Inter-Quartile Range); unit: papules and pustules] — The total number of papules and pustules on the patient was assessed.
  papules and pustules | 13.00 [7.33 to 44.67]
Clinician's Global Severity Score for Rosacea [Median (Inter-Quartile Range); unit: score on a scale] — Scale range: 0-4 (0=none to very mild; 1=mild; 2=moderate; 3=severe; 4=very severe).
  score on a scale | 1.83 [1.33 to 3.17]
Clinician's Global Erythema Assessment Score [Median (Inter-Quartile Range); unit: score on a scale] — Scale range: 0-4 (0=none; 1=mild; 2=moderate; 3=significant; 4=severe).
  score on a scale | 1.67 [1.17 to 3.00]
Rosacea Quality of Life (RosaQoL) Score [Median (Inter-Quartile Range); unit: score on a scale] — Scale range: 0-5 with greater scores denoting worse quality of life.
  score on a scale | 3.48 [2.57 to 4.24]
Immune Infiltrates in Papulopustular Rosacea Lesions [Median (Inter-Quartile Range); unit: score on a scale] — Immune infiltrates as assessed by immunohistochemistry, using a semi-quantitative grading scale for histological inflammation (scale range: 0-4, with 0-normal to 4-widespread inflammation).
  score on a scale | 2.50 [2.38 to 3.50]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Papule/Pustule Count at Week 16
Description: The total number of papules and pustules on the patient was assessed.
Time Frame: Baseline, week 16
Population: Participants who completed through week 16 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: papules and pustules
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 17
papules and pustules | -5.00 [-17.6 to 1.00]
Statistical Analysis 1: Comparison: Secukinumab Arm; The null hypothesis is that there would be no difference in papule/pustule count at baseline and after 16 weeks of secukinumab; the alternative hypothesis is that there would be a difference. Using an alpha=0.05 and power=0.80 (two sided test), the sample size needed would be 20. Assuming a dropout rate of 20%, 24 patients would be needed to achieve sufficient sample size; Test type: Other; p = 0.01, Wilcoxon signed rank test

2. Secondary Outcome: Change From Baseline Papule/Pustule Count at Week 12
Description: The total number of papules and pustules on the patient was assessed.
Time Frame: Baseline, week 12
Population: Participants who completed through week 12 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: papules and pustules
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 17
papules and pustules | -7.00 [-16.66 to 0.00]
Statistical Analysis 1: Comparison: Secukinumab Arm; Test type: Other; p = 0.02, Wilcoxon signed rank test

3. Secondary Outcome: Change From Baseline in Clinician's Global Severity Score for Rosacea at Week 16
Description: Scale range: 0-4 (0=none to very mild; 1=mild; 2=moderate; 3=severe; 4=very severe).
Time Frame: Baseline, week 16
Population: Participants who completed through week 16 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 17
score on a scale | -0.33 [-0.83 to 0.17]
Statistical Analysis 1: Comparison: Secukinumab Arm; Test type: Other; p = 0.03, Wilcoxon signed rank test

4. Secondary Outcome: Change From Baseline in Clinician's Global Erythema Assessment Score at Week 16
Description: Scale range: 0-4 (0=none; 1=mild; 2=moderate; 3=significant; 4=severe).
Time Frame: Baseline, week 16
Population: Participants who completed through week 16 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 17
score on a scale | -0.33 [-0.83 to 0.17]
Statistical Analysis 1: Comparison: Secukinumab Arm; Test type: Other; p = 0.2, Wilcoxon signed rank test

5. Secondary Outcome: Change From Baseline in Rosacea Quality of Life (RosaQoL) Score at Week 16
Description: Scale range: 0-5 with greater scores denoting worse quality of life.
Time Frame: Baseline, week 16
Population: Participants who completed through week 16 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 17
score on a scale | -0.61 [-1.53 to -0.14]
Statistical Analysis 1: Comparison: Secukinumab Arm; Test type: Other; p < 0.001, Wilcoxon signed rank test

6. Secondary Outcome: Count of Participants With ≥ Grade 3 Adverse Events
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 24
Participants | 0

7. Secondary Outcome: Change From Baseline in Immune Infiltrates in Papulopustular Rosacea Lesions at Week 16
Description: Immune infiltrates as assessed by immunohistochemistry, using a semi-quantitative grading scale for histological inflammation (scale range: 0-4, with 0-normal to 4-widespread inflammation).
Time Frame: Baseline, week 16
Population: Participants who contributed skin biopsies at both week 0 and week 16 are included in the analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Secukinumab Arm
Number analyzed (Participants) | 7
score on a scale | 0.43 [-0.25 to 1.50]
Statistical Analysis 1: Comparison: Secukinumab Arm; Test type: Other; p = 0.56, Wilcoxon signed rank test

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Secukinumab Arm
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 11/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab Arm (N=24)
Skin or nail infection (Infections and infestations) | 4
Otitis externa (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 3
Flu like symptoma (General disorders) | 1
Injection site reaction (General disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash (eczema) (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT03079531/Prot_SAP_000.pdf